CLINICAL TRIAL: NCT06615349
Title: DigiPall; a Randomized Controlled Trial of Digital Patient Reported Outcome and Biomarker Monitoring in Palliative Care
Brief Title: DigiPall; a Trial of Digital Patient Reported Outcome and Biomarker Monitoring in Palliative Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: David Blum (Other)
Collaborators: Zurich University of Applied Sciences (Other)
Responsible Party: Sponsor-Investigator, David Blum, Medical Director Palliative Care Center USZ, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: digiPall
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Terminal Illness; Terminal Cancer
Keywords: Palliative Care; chatbot; wearable; PROMs; rehospitalisation; mobile health

STUDY DESIGN:
Intervention Model Description: prospective, randomized, controlled
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DigiPall (Experimental): Patients receive standard of care + DigiPall intervention
  Interventions: Behavioral: DigiPall
- control (No Intervention): Patients receive standard of care

INTERVENTIONS:
Behavioral: DigiPall — DigiPall is an intervention combining a sensor-equipped wearable with a chatbot communicating via WhatsApp on the patient's smartphone. Patients will be asked two questions daily for their subjective rating through WhatsApp on their smartphone, worded slightly differently depending on the measured values for steps, heart rate and compliance as well as the patient's answer the day before.
  Arms: DigiPall

SUMMARY:
The aim of this study is to test if a system consisting of a wearable device measuring heartbeats and steps, together with daily communication with a chatbot on the smartphone asking the patients about their symptoms and giving tips, can reduce unplanned hospital readmissions and improve well-being in advanced cancer and severely ill patients.

DETAILED DESCRIPTION:
The aim of this study is to test the effect of a remote symptom and digital biomarker monitoring system on unplanned hospital readmissions, quality of life and sense of security in advanced cancer patients and patients with severe illnesses in palliative care.

Patients with cancer or other life-threatening illnesses are often burdened with pain and other distressing symptoms. Palliative care is an approach to prevent and relief suffering by means of early identification, assessment and treatment of these symptoms with the overall aim to improve quality of life of patients.

Palliative care wards are established in larger hospitals in Switzerland and provide short-term acute treatment of patients with incurable diseases. More than half of the patients are discharged home. However, unplanned rehospitalisations and emergency visits unfortunately occur frequently. Unplanned rehospitalisations are burdensome for the patient and caregiver and they are associated with higher costs. Up to 50% of unplanned rehospitalisations or hospital readmissions are deemed avoidable.

An unplanned hospital readmission within a specified time frame is an often applied quality benchmark in health care. When patients are discharged from specific palliative care wards, a good interprofessional outpatient or home care service has been most effective. However, close monitoring through home care teams is time consuming, costly, hindered by long distances and home care teams are not available everywhere. Furthermore, in many European countries primary care practices are rarified and reimbursement of home visits are insufficient. Therefore, new and innovative approaches for monitoring of this patient group are needed, especially in view of a growing number of patients and a decreasing number of care givers.

In the digital era self tracking is becoming more fashionable and daily screen-time is increasing. Concerning symptoms and well-being, patients monitoring themselves is the best option, because only they can adequately determine how they feel. Performance status and its deterioration can be remotely assessed by wearables. Mobile health technology is an easy and feasible way to monitor activity and health status.

This randomized controlled study aims to compare two groups of palliative patients, both receiving standard treatment with the intervention group additionally receiving the monitoring system. In the DigiPall intervention group, biomarker data is continuously gathered by a wearable device and questions about their subjective health status will be answered by the patients through chat. Based on their answers, automated feedback is provided. This feedback will not include any new prescriptions or suggest anything that was not already discussed with the treating physician, rather it will be reminding the patient of options in accordance to the existing treatment plan. There is strong evidence pointing to patients failing to implement the suggested treatment plan after discharge being a key factor in avoidable rehospitalisations. Therefore, the goal of the intervention is to strengthen the patient's self-management ability and sense of security, resulting in a better outcome in addition to reducing health care cost.

This approach has been well received in the feasibility study and the current study design has been developed with input by the patients themselves. During the study a patient group for advice will be consulted periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients with established diagnosis of a metastatic cancer/severe illness with limited life expectancy receiving palliative care services
* Estimated life expectancy <24 months (physician's guess)/ >3 months
* Karnofsky Index ≥ 50% / ECOG≤ 2
* Aged >18 years
* Owns and uses a smartphone
* Give written informed consent

Exclusion Criteria:

* Patients under curative treatment
* Relevant cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
rate of unplanned rehospitalisations and emergency visits | 84 days
  measure will be derived from hospital reports as well as statements by the patient on a weekly basis

SECONDARY OUTCOMES:
Quality of Life in palliative cancer care patients (EORTC QLQ-C15-PAL) | 91 days
  14 items scored from 1-4, higher score indicates worse outcome
  1 item scored from 1-7, higher score indicates better outcome
Sense of Security in Care - Patient Edition (SEC-P) | 91 days
  16 items scored from 1-6, higher score indicates better outcome
survival | 365 days
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: David Blum, MD PhD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wheatley VJ, Baker JI. "Please, I want to go home": ethical issues raised when considering choice of place of care in palliative care. Postgrad Med J. 2007 Oct;83(984):643-8. doi: 10.1136/pgmj.2007.058487. PMID 17916873
- [Background] Alsirafy SA, Raheem AA, Al-Zahrani AS, Mohammed AA, Sherisher MA, El-Kashif AT, Ghanem HM. Emergency Department Visits at the End of Life of Patients With Terminal Cancer: Pattern, Causes, and Avoidability. Am J Hosp Palliat Care. 2016 Aug;33(7):658-62. doi: 10.1177/1049909115581819. Epub 2015 Apr 15. PMID 25877944
- [Background] Donze JD, Lipsitz S, Schnipper JL. Risk Factors and Patterns of Potentially Avoidable Readmission in Patients With Cancer. J Oncol Pract. 2017 Jan;13(1):e68-e76. doi: 10.1200/JOP.2016.011445. Epub 2016 Oct 23. PMID 28084884
- [Background] Gerhardt G, Yemane A, Hickman P, Oelschlaeger A, Rollins E, Brennan N. Medicare readmission rates showed meaningful decline in 2012. Medicare Medicaid Res Rev. 2013 May 28;3(2):mmrr.003.02.b01. doi: 10.5600/mmrr.003.02.b01. eCollection 2013. PMID 24753966
- [Background] Chang VT, Hwang SS, Feuerman M, Kasimis BS. Symptom and quality of life survey of medical oncology patients at a veterans affairs medical center: a role for symptom assessment. Cancer. 2000 Mar 1;88(5):1175-83. doi: 10.1002/(sici)1097-0142(20000301)88:53.0.co;2-n. PMID 10699909
- [Background] Peters L, Sellick K. Quality of life of cancer patients receiving inpatient and home-based palliative care. J Adv Nurs. 2006 Mar;53(5):524-33. doi: 10.1111/j.1365-2648.2006.03754.x. PMID 16499673
- [Background] LeBlanc TW, Nickolich M, Rushing CN, Samsa GP, Locke SC, Abernethy AP. What bothers lung cancer patients the most? A prospective, longitudinal electronic patient-reported outcomes study in advanced non-small cell lung cancer. Support Care Cancer. 2015 Dec;23(12):3455-63. doi: 10.1007/s00520-015-2699-4. Epub 2015 Mar 21. PMID 25791391
- [Background] Delgado-Guay MO, Rodriguez-Nunez A, Shin SH, Chisholm G, Williams J, Frisbee-Hume S, Bruera E. Characteristics and outcomes of patients with advanced cancer evaluated by a palliative care team at an emergency center. A retrospective study. Support Care Cancer. 2016 May;24(5):2287-2295. doi: 10.1007/s00520-015-3034-9. Epub 2015 Nov 21. PMID 26590844
- [Background] Tsai SC, Liu LN, Tang ST, Chen JC, Chen ML. Cancer pain as the presenting problem in emergency departments: incidence and related factors. Support Care Cancer. 2010 Jan;18(1):57-65. doi: 10.1007/s00520-009-0630-6. Epub 2009 Apr 7. PMID 19350283
- [Background] Elsayem AF, Elzubeir HE, Brock PA, Todd KH. Integrating palliative care in oncologic emergency departments: Challenges and opportunities. World J Clin Oncol. 2016 Apr 10;7(2):227-33. doi: 10.5306/wjco.v7.i2.227. PMID 27081645
- [Background] Delgado-Guay MO, Kim YJ, Shin SH, Chisholm G, Williams J, Allo J, Bruera E. Avoidable and unavoidable visits to the emergency department among patients with advanced cancer receiving outpatient palliative care. J Pain Symptom Manage. 2015 Mar;49(3):497-504. doi: 10.1016/j.jpainsymman.2014.07.007. Epub 2014 Aug 15. PMID 25131891
- [Background] Henson LA, Gao W, Higginson IJ, Smith M, Davies JM, Ellis-Smith C, Daveson BA. Emergency department attendance by patients with cancer in their last month of life: a systematic review and meta-analysis. J Clin Oncol. 2015 Feb 1;33(4):370-6. doi: 10.1200/JCO.2014.57.3568. Epub 2014 Dec 22. PMID 25534384
- [Background] Witt D, Kellogg R, Snyder M, Dunn J. Windows Into Human Health Through Wearables Data Analytics. Curr Opin Biomed Eng. 2019 Mar;9:28-46. doi: 10.1016/j.cobme.2019.01.001. Epub 2019 Jan 28. PMID 31832566
- [Background] Urrea B, Misra S, Plante TB, Kelli HM, Misra S, Blaha MJ, Martin SS. Mobile Health Initiatives to Improve Outcomes in Primary Prevention of Cardiovascular Disease. Curr Treat Options Cardiovasc Med. 2015 Dec;17(12):59. doi: 10.1007/s11936-015-0417-7. PMID 26474892
- [Background] Mendoza M, Han M, Meyring-Wosten A, Wilund K, Kotanko P. It's a non-dialysis day... Do you know how your patient is doing? A case for research into interdialytic activity. Blood Purif. 2015;39(1-3):74-83. doi: 10.1159/000369430. Epub 2015 Jan 20. PMID 25662096
- [Background] Strohrmann C, Labruyere R, Gerber CN, van Hedel HJ, Arnrich B, Troster G. Monitoring motor capacity changes of children during rehabilitation using body-worn sensors. J Neuroeng Rehabil. 2013 Jul 30;10:83. doi: 10.1186/1743-0003-10-83. PMID 23899401
- [Background] Seiter J, Derungs A, Schuster-Amft C, Amft O, Troster G. Daily life activity routine discovery in hemiparetic rehabilitation patients using topic models. Methods Inf Med. 2015;54(3):248-55. doi: 10.3414/ME14-01-0082. Epub 2015 Feb 6. PMID 25658903
- [Background] Muaremi A, Arnrich B, Troster G. Towards Measuring Stress with Smartphones and Wearable Devices During Workday and Sleep. Bionanoscience. 2013;3(2):172-183. doi: 10.1007/s12668-013-0089-2. PMID 25530929
- [Background] Bennett AV, Jensen RE, Basch E. Electronic patient-reported outcome systems in oncology clinical practice. CA Cancer J Clin. 2012 Sep-Oct;62(5):337-47. doi: 10.3322/caac.21150. Epub 2012 Jul 18. PMID 22811342
- [Background] Brunelli C, Kaasa S, Knudsen AK, Hjermstad MJ, Pigni A, Caraceni A. Comparisons of patient and physician assessment of pain-related domains in cancer pain classification: results from a large international multicenter study. J Pain. 2014 Jan;15(1):59-67. doi: 10.1016/j.jpain.2013.09.011. Epub 2013 Oct 2. PMID 24373570
- [Background] Lundstrom S. Is it reliable to use cellular phones for symptom assessment in palliative care? Report on a study in patients with advanced cancer. J Palliat Med. 2009 Dec;12(12):1087. doi: 10.1089/jpm.2009.0207. No abstract available. PMID 19995287
- [Background] Basch E, Deal AM, Dueck AC, Scher HI, Kris MG, Hudis C, Schrag D. Overall Survival Results of a Trial Assessing Patient-Reported Outcomes for Symptom Monitoring During Routine Cancer Treatment. JAMA. 2017 Jul 11;318(2):197-198. doi: 10.1001/jama.2017.7156. PMID 28586821
- [Background] Ferriolli E, Skipworth RJ, Hendry P, Scott A, Stensteth J, Dahele M, Wall L, Greig C, Fallon M, Strasser F, Preston T, Fearon KC. Physical activity monitoring: a responsive and meaningful patient-centered outcome for surgery, chemotherapy, or radiotherapy? J Pain Symptom Manage. 2012 Jun;43(6):1025-35. doi: 10.1016/j.jpainsymman.2011.06.013. Epub 2012 Jan 24. PMID 22269181
- [Background] Kaasa S, Loge JH, Fayers P, Caraceni A, Strasser F, Hjermstad MJ, Higginson I, Radbruch L, Haugen DF. Symptom assessment in palliative care: a need for international collaboration. J Clin Oncol. 2008 Aug 10;26(23):3867-73. doi: 10.1200/JCO.2007.15.8881. PMID 18688054
- [Background] Abernethy AP, Currow DC. Patient self-reporting in palliative care using information technology: Yes, there is hope! Palliat Med. 2011 Oct;25(7):673-4. doi: 10.1177/0269216311422760. No abstract available. PMID 21987664
- [Background] Cox A, Illsley M, Knibb W, Lucas C, O'Driscoll M, Potter C, Flowerday A, Faithfull S. The acceptability of e-technology to monitor and assess patient symptoms following palliative radiotherapy for lung cancer. Palliat Med. 2011 Oct;25(7):675-81. doi: 10.1177/0269216311399489. Epub 2011 Apr 7. PMID 21474620
- [Background] Skipworth RJ, Stene GB, Dahele M, Hendry PO, Small AC, Blum D, Kaasa S, Trottenberg P, Radbruch L, Strasser F, Preston T, Fearon KC, Helbostad JL; European Palliative Care Research Collaborative (EPCRC). Patient-focused endpoints in advanced cancer: criterion-based validation of accelerometer-based activity monitoring. Clin Nutr. 2011 Dec;30(6):812-21. doi: 10.1016/j.clnu.2011.05.010. Epub 2011 Jul 5. PMID 21733604
- [Background] Ng A, Gupta E, Bansal S, Fontillas RC, Amos CE Jr, Williams JL, Dibaj S, Bruera E. Cancer Patients' Perception of Usefulness of Wearable Exercise Trackers. PM R. 2021 Aug;13(8):845-851. doi: 10.1002/pmrj.12475. Epub 2020 Oct 20. PMID 32844592
- [Background] Pavic M, Klaas V, Theile G, Kraft J, Troster G, Blum D, Guckenberger M. Mobile Health Technologies for Continuous Monitoring of Cancer Patients in Palliative Care Aiming to Predict Health Status Deterioration: A Feasibility Study. J Palliat Med. 2020 May;23(5):678-685. doi: 10.1089/jpm.2019.0342. Epub 2019 Dec 23. PMID 31873052
- [Background] Blum D, Koeberle D, Omlin A, Walker J, Von Moos R, Mingrone W, deWolf-Linder S, Hayoz S, Kaasa S, Strasser F, Ribi K. Feasibility and acceptance of electronic monitoring of symptoms and syndromes using a handheld computer in patients with advanced cancer in daily oncology practice. Support Care Cancer. 2014 Sep;22(9):2425-34. doi: 10.1007/s00520-014-2201-8. Epub 2014 Apr 5. PMID 24705855
- [Background] Blum D, Koeberle D, Ribi K, Schmitz SF, Utiger U, Klingbiel D, Strasser F. Electronic monitoring of symptoms and syndromes associated with cancer: methods of a randomized controlled trial SAKK 95/06 E-MOSAIC. BMC Palliat Care. 2012 Sep 24;11:19. doi: 10.1186/1472-684X-11-19. PMID 23006802
- [Background] Strasser F, Blum D, von Moos R, Cathomas R, Ribi K, Aebi S, Betticher D, Hayoz S, Klingbiel D, Brauchli P, Haefner M, Mauri S, Kaasa S, Koeberle D; Swiss Group for Clinical Cancer Research (SAKK). The effect of real-time electronic monitoring of patient-reported symptoms and clinical syndromes in outpatient workflow of medical oncologists: E-MOSAIC, a multicenter cluster-randomized phase III study (SAKK 95/06). Ann Oncol. 2016 Feb;27(2):324-32. doi: 10.1093/annonc/mdv576. Epub 2015 Dec 8. PMID 26646758
- [Background] Calvert M, Kyte D, Mercieca-Bebber R, Slade A, Chan AW, King MT; the SPIRIT-PRO Group; Hunn A, Bottomley A, Regnault A, Chan AW, Ells C, O'Connor D, Revicki D, Patrick D, Altman D, Basch E, Velikova G, Price G, Draper H, Blazeby J, Scott J, Coast J, Norquist J, Brown J, Haywood K, Johnson LL, Campbell L, Frank L, von Hildebrand M, Brundage M, Palmer M, Kluetz P, Stephens R, Golub RM, Mitchell S, Groves T. Guidelines for Inclusion of Patient-Reported Outcomes in Clinical Trial Protocols: The SPIRIT-PRO Extension. JAMA. 2018 Feb 6;319(5):483-494. doi: 10.1001/jama.2017.21903. PMID 29411037
- [Background] Groenvold M, Petersen MA, Aaronson NK, Arraras JI, Blazeby JM, Bottomley A, Fayers PM, de Graeff A, Hammerlid E, Kaasa S, Sprangers MA, Bjorner JB; EORTC Quality of Life Group. The development of the EORTC QLQ-C15-PAL: a shortened questionnaire for cancer patients in palliative care. Eur J Cancer. 2006 Jan;42(1):55-64. doi: 10.1016/j.ejca.2005.06.022. Epub 2005 Sep 12. PMID 16162404
- [Background] Basch E, Deal AM, Kris MG, Scher HI, Hudis CA, Sabbatini P, Rogak L, Bennett AV, Dueck AC, Atkinson TM, Chou JF, Dulko D, Sit L, Barz A, Novotny P, Fruscione M, Sloan JA, Schrag D. Symptom Monitoring With Patient-Reported Outcomes During Routine Cancer Treatment: A Randomized Controlled Trial. J Clin Oncol. 2016 Feb 20;34(6):557-65. doi: 10.1200/JCO.2015.63.0830. Epub 2015 Dec 7. PMID 26644527
- [Background] Hamine S, Gerth-Guyette E, Faulx D, Green BB, Ginsburg AS. Impact of mHealth chronic disease management on treatment adherence and patient outcomes: a systematic review. J Med Internet Res. 2015 Feb 24;17(2):e52. doi: 10.2196/jmir.3951. PMID 25803266
- [Background] Bradley EH, Curry L, Horwitz LI, Sipsma H, Thompson JW, Elma M, Walsh MN, Krumholz HM. Contemporary evidence about hospital strategies for reducing 30-day readmissions: a national study. J Am Coll Cardiol. 2012 Aug 14;60(7):607-14. doi: 10.1016/j.jacc.2012.03.067. Epub 2012 Jul 18. PMID 22818070
- [Background] Krevers B, Milberg A. The instrument 'sense of security in care--patients' evaluation': its development and presentation. Psychooncology. 2014 Aug;23(8):914-20. doi: 10.1002/pon.3502. Epub 2014 Feb 14. PMID 24677414
- [Background] Wallace EM, Cooney MC, Walsh J, Conroy M, Twomey F. Why do palliative care patients present to the emergency department? Avoidable or unavoidable? Am J Hosp Palliat Care. 2013 May;30(3):253-6. doi: 10.1177/1049909112447285. Epub 2012 May 23. PMID 22628898